CLINICAL TRIAL: NCT05164679
Title: A Feasibility Study of Training in a Local Community Aimed Upon Health Promotion With Special Emphasis on Musculoskeletal Health Effects
Brief Title: Training in a Local Community Aimed Upon Musculoskeletal Health Promotion for Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ewa Wulff Helge, Associate Professor, Ph.D., University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Knoglestaerk
Record Dates: First submitted 2021-12-04; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Age-Related Osteoporosis
Keywords: Bone mineral density; bone turnover marker; high-impact; odd-impact; resistance exercise; menopause; health promotion
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: Healthy, sedentary postmenopausal women aged below 70 years were eligible to participate in the present study.
  Inclusion criteria were:
  * non-smoker
  * body mass index (BMI) <30 kg/m2.
  Exclusion criteria were:
  * T-score < -3 SD in the lumbar spine or hip
  * high BMD in relation to age (Z-score > 1.5 SD)
  * use of hormone therapy, medical treatment, or supplements that affect bone metabolism
  * previous or current medical condition affecting bone health
  * engagement in regular and systematic weight-bearing training or strength training during the preceding two years.
  Initially, twenty women were recruited to the training via an online advertisement and a local newspaper, but only 19 showed up for pre-testing. After a medical examination, one participant was excluded due to low BMD (T-score < -3 SD), and two were excluded due to high BMI (≥30 kg/m2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMT (Experimental): Intervention group performing multimodal training (MMT) 1-2 hours weekly
  Interventions: Behavioral: multimodal training (MMT)
- CON (No Intervention): Sedentary control group

INTERVENTIONS:
Behavioral: multimodal training (MMT) — Supervised multimodal exercise training (MMT) performed 1-2 hours weekly for 19 weeks
  Other Names: Sedentary control group (CON)
  Arms: MMT

SUMMARY:
To minimize fracture risk, diverse and varied training of high intensity (multimodal training) is recommended to increase bone strength. However, the effectiveness of different training programmes performed in community settings remain uncertain. The present study aimed to evaluate the feasibility and the effectiveness of 19-week of multimodal training in a local community center in Copenhagen, Denmark. The health promotion initiative had special emphasis on musculoskeletal health in postmenopausal women.

DETAILED DESCRIPTION:
A local community center was offering supervised multimodal training (MMT) to postmenopausal, healthy women twice weekly, and the aim of the present study was to evaluate the feasibility and the musculoskeletal health promoting effects of the training. The evaluation study lasted for 19 weeks, and the average attendance rate of MMT participants had to be > 1 hour weekly. The primary outcomes were bone mineral density (BMD) assessed by Dual-Energy X-ray Absorptiometry (DXA) scanning and the fasted plasma concentration of bone turnover markers (BTM): N-terminal propeptide of type I procollagen (P1NP) , C-terminal telopeptide of type I collagen (CTX), Osteocalcin), while secondary outcomes were body composition variables, dynamic postural balance and functional muscle strength. To test within- and between-group differences in the pre and post outcomes the training group (MMT) was compared with a sedentary control group (CON).

Every participant was fully informed before giving her written informed consent to the procedures and potential discomfort associated with the study. The study was conducted in accordance with the Declaration of Helsinki and approved by the local ethics committee of the Capital Region of Denmark, H-18044190.

ELIGIBILITY:
Inclusion Criteria:

* past menopause
* non-smoking
* BMI <30 kg/m2

Exclusion Criteria:

* T-score < -3 SD in the lumbar spine or hip
* Z-score > 1.5 SD)
* use of hormone therapy, medical treatment or supplements that affect bone metabolism
* previous or current medical condition affecting bone health
* engagement in regular and systemic weight-bearing training or strength training during the preceding two years

Max Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Whole-body and regional BMD | 19 weeks
  bone mineral density (g/cm2)
Osteocalcin | 3 weeks and 19 weeks
  Concentration of Osteocalcin in plasma in fasted state (µg/l)
P1NP | 3 weeks and 19 weeks
  Concentration of P1NP in plasma in fasted state (µg/l)
CTX | 3 weeks and 19 weeks
  Concentration of CTX in plasma in fasted state (ng/l)

SECONDARY OUTCOMES:
Body fat percentage | 19 weeks
  Body fat percentage (%)
Visceral adipose tissue (VAT) | 19 weeks
  Volume (m3)
Body weight | 19 weeks
  kg
BMI | 19 weeks
  kg/m2
Total fat mass | 19 weeks
  kg
Total lean body mass (LBM) | 19 weeks
  kg
Whole-body bone mineral content (BMC) | 19 weeks
  g
dynamic balance | 19 weeks
  time to fulfill a four-square-balance test (sec)
dynamic muscle strength | 19 weeks
  Jump-and-reach-test (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Eva W Helge, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

REFERENCES:
- [Derived] Prawiradilaga RS, Bendtsen M, Esrup S, Jorgensen NR, Yulianto FA, Helge EW. Feasibility Study of Community-Based Training for Musculoskeletal Health Promotion. F1000Res. 2024 Sep 4;11:51. doi: 10.12688/f1000research.73698.3. eCollection 2022. PMID 39263388

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05164679/Prot_SAP_000.pdf